CLINICAL TRIAL: NCT06046443
Title: A Randomized, Placebo-controlled, Double-Blind Phase 2 Study to Assess Efficacy and Safety of LB54640 in Patients With Hypothalamic Obesity, With an Open-Label Extension
Brief Title: A Study to Assess Efficacy and Safety of LB54640 in Patients With Hypothalamic Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LG-MCCL005
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypothalamic Obesity
Keywords: melanocortin 4 receptor, MC4R; MC4R agonism
MeSH Terms: conditions — Sexual Infantilism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LB54640 Low dose (Experimental): Participants will be randomized to receive LB54640 low dose, middle dose, or high dose, or placebo by oral administration in a 1:1:1:1 ratio.
  Interventions: Drug: LB54640
- LB54640 Middle dose (Experimental): Participants will be randomized to receive LB54640 low dose, middle dose, or high dose, or placebo by oral administration in a 1:1:1:1 ratio.
  Interventions: Drug: LB54640
- LB54640 High dose (Experimental): Participants will be randomized to receive LB54640 low dose, middle dose, or high dose, or placebo by oral administration in a 1:1:1:1 ratio.
  Interventions: Drug: LB54640
- Placebo (Placebo Comparator): Participants will be randomized to receive LB54640 low dose, middle dose, or high dose, or placebo by oral administration in a 1:1:1:1 ratio.
  Interventions: Drug: Placebo
- Open-label LB54640 (Experimental): Eligible participants who provide consent to continue into the open-label portion of the study will receive open-label LB54640.
  Interventions: Drug: LB54640

INTERVENTIONS:
Drug: LB54640 — Oral daily administration
  Arms: LB54640 High dose; LB54640 Low dose; LB54640 Middle dose; Open-label LB54640
Drug: Placebo — Placebo matched to LB54640
  Arms: Placebo

SUMMARY:
The goal of this study is to determine how well LB54640 works and how safe it is in patients with Hypothalamic Obesity (HO). The study will evaluate the effect of LB54640 on safety, weight reduction, hunger, and quality of life in patients 12 years of age and older with HO. Patients will take an oral daily dose of either LB54640 (low, middle, or high dose) or placebo through Week 14. Eligible patients who consent to continue in the study after Week 14 will take an oral daily dose of LB54640 through Week 56.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented evidence of acquired hypothalamic obesity (HO)
* Age 12 years and older
* Weight gain associated with the hypothalamic injury and a BMI of ≥30 kg/m2 for patients ≥18 years of age or BMI ≥95th percentile for age and sex for patients <18 years of age
* Male and female participants agree to follow study contraception requirements and use a highly effective form of contraception throughout the study and for 90 days after the study

Key Exclusion Criteria:

* Weight loss >2% in the previous 3 months for patients ≥18 years of age or >2% reduction in BMI for patients <18 years of age
* History of major surgical procedure within 30 days
* HbA1c >10.9%
* Fasting glucose level >270 mg/dL
* Previous use of MC4R agonists
* Diagnosis of Prader-Willi syndrome (PWS) or Rapid-onset obesity with hypoventilation, hypothalamic, autonomic dysregulation, neuroendocrine tumor syndrome (ROHHADNET).
* Diagnosis of severe psychiatric disorders; any suicidal ideation, attempt or behavior
* History or close family history of skin cancer or melanoma
* Current clinically significant pulmonary, cardiac, or oncologic disease considered severe enough to interfere with the study and/or confound the results

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-02-09 (Actual); Study Completion 2026-02-09 (Actual)

PRIMARY OUTCOMES:
Mean percentage change in BMI | From Baseline to Week 14

SECONDARY OUTCOMES:
Frequency and severity of adverse events (AEs) | From Baseline to Week 52
Mean change in BMI | Baseline to Weeks 6, 10, 14
Proportion of patients who achieve ≥5% reduction in body weight | Baseline to Week 14
Mean change in the weekly average of the daily most hunger score | Baseline to Week 14
Mean change and mean percentage change from baseline in body weight | From Baseline to Week 52
Mean change and mean percentage change from baseline in waist circumference. | From Baseline to Week 52
Mean change and mean percentage change from baseline in body composition assessed by dual energy x-ray absorptiometry | From Baseline to Week 52
  Fat mass and lean mass will be measured through dual energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (10):
- United States (7):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- United Kingdom (3):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - University of Cambridge, Cambridge
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No